CLINICAL TRIAL: NCT00407134
Title: Acute Haemodynamic Effects of Peritoneal Dialysis as Evaluated by Sphygmocor Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/382
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Different abdominal volumes and different glucose-concentrations during peritoneal dialysis

SUMMARY:
Subjects with peritoneal dialysis are randomized to different groups. The different groups receive different intra-abdominal volumes and different glucose-concentrations.

The effects on blood pressure and other cardiovascular parameters (e.g. central blood pressure, augmentation index, ...) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with peritoneal dialysis
* Aged 18-80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be